CLINICAL TRIAL: NCT02104752
Title: Curcumin as a Novel Treatment to Improve Cognitive Dysfunction in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: Stanley Medical Research Institute (Other); Theravalues, Inc. (Industry); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael C. Davis, M.D., Ph.D., Physician, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-121701
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Cognition; Psychosis
Keywords: Curcumin; Turmeric; Schizophrenia; Cognition; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin (Experimental): Curcumin capsules (Theracurmin formulation of curcumin nanoparticles). Subjects randomized to curcumin will receive 360 mg/day (divided into twice daily oral doses).
  Interventions: Drug: Curcumin
- Sugar Pill (Placebo Comparator): Matched placebo, 2 capsules twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — 360 mg/day (divided into twice daily oral doses)
  Other Names: Theracurmin; Curcumin nanoparticles
  Arms: Curcumin
Drug: Placebo — Inactive, matched placebo ("Sugar Pill")
  Arms: Sugar Pill

SUMMARY:
The investigators propose to test whether curcumin nanoparticles will improve behavioral measures and biomarkers of cognition and neuroplasticity in patients with schizophrenia who are already receiving a stable dose of antipsychotic.

DETAILED DESCRIPTION:
The investigators will use a formulation of curcumin with high bioavailability that possesses a pharmacokinetic profile expected to exert biological effects. Specifically, 36 subjects will be enrolled in the double-blind randomized controlled trial. They will be randomized to curcumin or placebo for 8 weeks. At baseline, and 4 and 8 weeks, subjects will receive assessments of neurocognition (e.g., processing speed, attention and vigilance, working memory, learning, reasoning and problem solving), social cognition, EEG biomarkers (e.g., visual cortical plasticity and mismatch negativity), a serum marker of neurogenesis (BDNF levels), and clinical symptoms (positive and negative symptoms). At weeks 2 and 6 subjects will return for additional safety (e.g., vitals, side effects, akathisia) and medication adherence assessments. Improvement on the primary outcome measure (MATRICS Consensus Cognitive Battery), as well as secondary outcome measures, will be compared between participants randomized to placebo versus curcumin. The results of this study will establish whether curcumin is a viable adjunctive agent for future larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia
* age 18 - 65 years
* understand spoken English sufficiently to comprehend testing procedures
* corrected vision of at least 20/30
* currently prescribed an antipsychotic medication

Exclusion Criteria:

* clinically significant neurological disease determined by medical history (e.g., epilepsy)
* history of serious head injury (i.e., loss of consciousness > 1 hr., no neuropsychological sequelae, no cognitive rehabilitation post head injury)
* sedatives or benzodiazepines within 12 hrs of testing
* any psychiatric hospitalization within 3 months prior to study participation
* behaviors suggesting any potential danger to self or others within 6 months prior to study participation
* antipsychotic dose change more than 50% over the 3 months prior to study participation
* acute medical problems or untreated chronic medical conditions within 3 months prior to study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marder, M.D., Principal Investigator — VA Greater Los Angeles; Jonathan K Wynn, Ph.D., Principal Investigator — VA Greater Los Angeles; Michael C Davis, M.D.,Ph.D., Principal Investigator — VA Greater Los Angeles
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Hurley LL, Akinfiresoye L, Nwulia E, Kamiya A, Kulkarni AA, Tizabi Y. Antidepressant-like effects of curcumin in WKY rat model of depression is associated with an increase in hippocampal BDNF. Behav Brain Res. 2013 Feb 15;239:27-30. doi: 10.1016/j.bbr.2012.10.049. Epub 2012 Nov 8. PMID 23142609
- [Background] Dong S, Zeng Q, Mitchell ES, Xiu J, Duan Y, Li C, Tiwari JK, Hu Y, Cao X, Zhao Z. Curcumin enhances neurogenesis and cognition in aged rats: implications for transcriptional interactions related to growth and synaptic plasticity. PLoS One. 2012;7(2):e31211. doi: 10.1371/journal.pone.0031211. Epub 2012 Feb 16. PMID 22359574
- [Background] Sasaki H, Sunagawa Y, Takahashi K, Imaizumi A, Fukuda H, Hashimoto T, Wada H, Katanasaka Y, Kakeya H, Fujita M, Hasegawa K, Morimoto T. Innovative preparation of curcumin for improved oral bioavailability. Biol Pharm Bull. 2011;34(5):660-5. doi: 10.1248/bpb.34.660. PMID 21532153
- [Background] Shamsi S, Lau A, Lencz T, Burdick KE, DeRosse P, Brenner R, Lindenmayer JP, Malhotra AK. Cognitive and symptomatic predictors of functional disability in schizophrenia. Schizophr Res. 2011 Mar;126(1-3):257-64. doi: 10.1016/j.schres.2010.08.007. Epub 2010 Sep 15. PMID 20828991
- [Derived] Wynn JK, Green MF, Hellemann G, Karunaratne K, Davis MC, Marder SR. The effects of curcumin on brain-derived neurotrophic factor and cognition in schizophrenia: A randomized controlled study. Schizophr Res. 2018 May;195:572-573. doi: 10.1016/j.schres.2017.09.046. Epub 2017 Sep 29. No abstract available. PMID 28965778

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Curcumin | Sugar Pill
Started | 18 | 21
Completed | 17 | 19
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Weight gain; unrelated anxiety | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Sugar Pill | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.6) | 50.9 (10.6) | 50.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 11 | 19 | 30
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: This battery was developed as part of the National Institute of Mental Health (NIMH) sponsored Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Initiative to assess cognition in clinical trials of cognition enhancing drugs. The MCCB comprises 10 tests that assess 7 cognitive domains (speed of processing, verbal memory, visual memory, working memory, reasoning and problem solving, attention/vigilance, and social cognition). The MCCB takes approximately 65 minutes to administer and provides age and gender-corrected normed T-scores, including a global composite score and cognitive domain scores. The range of T-scores is between 0 to 100 with a mean of 50. Higher scores indicate better overall cognitive functioning.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Curcumin | Sugar Pill
Number analyzed (Participants) | 17 | 19
Score on a Scale
  Baseline | 36.6 (15.1) | 32.9 (10.3)
  Week 4 | 36.3 (14.5) | 33.8 (11.0)
  Week 8 | 35.8 (14.5) | 33.9 (9.7)

2. Secondary Outcome: Electroencephalogram (EEG) Mismatch Negativity Paradigm (MMN)
Description: A passive attention auditory oddball paradigm will be used to assess MMN. For MMN, difference waves generated by subtracting the standard from deviant event related potentials (ERP) will be analyzed. The specific electrodes used to examine each component will be chosen based on maximal activity seen by inspection of the topographical maps. More negative values indicate a larger (i.e., better) MMN response.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: microVolts
Arm/Group | Curcumin | Sugar Pill
Number analyzed (Participants) | 17 | 19
microVolts
  Baseline | -2.2 (2.16) | -1.84 (1.42)
  Week 4 | -2.15 (1.47) | -1.99 (1.84)
  Week 8 | -2.15 (1.66) | -1.68 (1.10)

3. Secondary Outcome: Brain Derived Neurotrophic Factor (BDNF)
Description: Serum will be collected at baseline, 4 weeks, and 8 weeks. BDNF concentrations will be quantified by enzyme-linked immunosorbent assay.
Time Frame: Baseline, Week 4, Week 8
Population: Participant dropped at the 8 week follow-up
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Curcumin | Sugar Pill
Number analyzed (Participants) | 17 | 19
pg/mL
  Baseline | 11416 (10067) | 14227 (9371)
  Week 4 | 15395 (11065) | 13288 (10565)
  Week 8: number analyzed (Participants) | 17 | 18
  Week 8 | 14828 (12876) | 10219 (8571)

4. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The Brief Psychiatric Rating Scale (BPRS) will be the primary measure for assessing positive symptoms. We will be using the UCLA expanded 24-item version of the scale. The total score ranges from 24-168, with lower scores being better (i.e., less symptomatology).
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Curcumin | Sugar Pill
Number analyzed (Participants) | 17 | 19
Score on a Scale
  Baseline | 36.1 (7.7) | 38.1 (9.5)
  Week 4 | 35.1 (5.7) | 37.9 (10.9)
  Week 8 | 36.1 (8.8) | 37.1 (10.7)

5. Secondary Outcome: The Clinical Assessment Interview for Negative Symptoms (CAINS)
Description: The Clinical Assessment Interview for Negative Symptoms (CAINS) will be used to assess negative symptoms. This scale is comprised of 9 items that rate motivation and pleasure symptoms and 4 items that rate expression symptoms.
  We are reporting the motivation subscale. The total score can range from 0-36 (summed over the 9 items), with lower scores being better (i.e., less symptomatology).
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Curcumin | Sugar Pill
Number analyzed (Participants) | 17 | 19
Score on a Scale
  Baseline | 14.2 (6.8) | 16.0 (5.9)
  Week 4 | 15.8 (7.5) | 16.2 (7.1)
  Week 8 | 15.1 (6.2) | 17.9 (7.8)

ADVERSE EVENTS:
Arm/Group | Curcumin | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No